CLINICAL TRIAL: NCT01703390
Title: Pilot Study: Biomarker Directed Treatment in Metastatic Colorectal Cancer
Brief Title: Biomarker Directed Treatment in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_ERCC1; 2011-003217-41 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; mCRC; ERCC-1; ERCC1; AGMT
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERCC-1 low (Experimental): modifiedFOLFOX6 + Cetuximab oxaliplatin 85 mg/m2 on day 1, 15 q d29 for 6 cycles folinic acid (FA) 400 mg/m2 on days 1 and 15 and q d29 for 6 cycles fluorouracil (5-FU) 400 mg/m2 bolus day 1 + 2400 mg/m2 46-hour infusion on days 1, 2 and 15, 16 and q d29 for 6 cycles or until unacceptable toxicity Cetuximab will be administered as a 120- minute intravenous infusion at 500 mg/m2 on day 1 then 500 mg/m2 bi-weekly
  Interventions: Drug: modifiedFOLFOX6 + Cetuximab
- ERCC-1 high (Experimental): FOLFIRI + Cetuximab irinotecan 180 mg/m² on day 1, 15 q d29 for 6 cycles folinic acid (FA)400 mg/m2 on days 1 and 15 and q d29 for 6 cycles fluorouracil (5-FU) 400 mg/m2 bolus + 2400 mg/m2 46-hour infusion on days 1, 2 and 15, 16 and q d29 for 6 cycles or until unacceptable toxicity Cetuximab will be administered as a 120- minute intravenous infusion at 500 mg/m2 on day 1 then 500 mg/m2 bi-weekly
  Interventions: Drug: FOLFIRI + Cetuximab

INTERVENTIONS:
Drug: FOLFIRI + Cetuximab
  Arms: ERCC-1 high
Drug: modifiedFOLFOX6 + Cetuximab
  Arms: ERCC-1 low

SUMMARY:
This pilot study is being mounted to assess whether treatment assignment by ERCC-1 gene expression status suggests better clinical results from historical experience in metastatic colorectal cancer (mCRC). In wild type KRAS mCRC patients treated with either FOLFOX or FOLFIRI in combination with cetuximab the median response rate is approximately 60-65%. Biomarker directed treatment in this study may demonstrate that patients with low ERCC-1 treated with FOLFOX and cetuximab, and those with high ERCC-1 treated with FOLFIRI and cetuximab, will improve response rate to 70-75%. KRAS wild type patients will be treated with 6 cycles of one of the following regimens chosen for optimization based on patient characteristics (primary treatment phase). Patients with ERCC-1 < 1.7 relative gene expression of ERCC-1 over ß-actin (ERCC-1 low) will be assigned to treatment with mFOLFOX6 in combination with Cetuximab. Patients with ERCC-1 gene expression > 1.7 relative gene expression of ERCC-1 over over ß-actin (ERCC-1 high) will be assigned to treatment with FOLFIRI in combination with Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

1.1 Inclusion criteria for pre-screening phase:

* Untreated advanced metastatic colorectal cancer patients
* Adequate tissue to evaluate for genotyping (10 x 10µm thick formalin fixed paraffin embedded tissue sections and one corresponding HE stained slide or a FFPE tumor block)

1.2 Inclusion criteria for treatment phase:

Patients must fulfill all criteria listed below prior to enrolment in the study:

* Untreated wild-type KRAS metastatic colorectal cancer
* Previous adjuvant therapy must have been completed > 6 months before therapy initiation on this study
* Age >18 years
* Measureable disease with CT or MRI
* ECOG performance status of 0-2
* Adequate organ function

  * Hematologic:

    * Absolute neutrophil count > 1,500/µL
    * Hemoglobin >9 mg/dl
    * Platelet count >100,000 /µl
  * Renal:

    * Serum creatinine <1.5 x Upper limit of normal (UPN) or estimated clearance > 30 ml/min
  * Hepatic:

    * Serum bilirubin < 1.5 mg/dl

Exclusion Criteria:

* Creatinine clearance below 30 ml/min
* Patients with a history of other malignancies within 2 years prior to study entry, except for adequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low grade, early stage localized prostate cancer treated surgically with curative intent; good prognosis DCIS of the breast treated with lumpectomy alone with curative intent.
* Patients with a history of severe cardiac disease; e.g. NYHA Functional Class III or IV heart failure, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, or unstable angina.
* Other known co-morbidity with the potential to dominate survival
* Hypersensitivity with anaphylactic reaction to humanized monoclonal antibodies or any of the applied drugs
* Pregnant or breast feeding women
* Any co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Response | 5 years
  Treatment response according to Response Evaluation Criteria In Solid Tumors [RECIST]

SECONDARY OUTCOMES:
Progression free survival (PFS) | 5 years
Response rate | 5 years
  Description of group differences between ERCC-1 low and ERCC-1 high patients with respect to response rate, PFS and OS
Patient characteristics | 5 years
  Description of group differences between ERCC-1 low and ERCC-1 high patients with respect to KRAS status
Secondary resection rate | 5 years
Molecular markers for toxicity | 5 years
Number of adverse events during study treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Winder, MD, Principal Investigator — LKH Feldkirch, Interne E
Locations (11):
- Austria (11):
  - A.ö. Bezirkskrankenhaus Kufstein, Innere Medizin / Hämatologie / Onkologie, Kufstein, Tyrol
  - KUK Linz - Med Campus III.: Univ.-Klinik für Hämatologie und Internistische Onkologie, Linz, Upper Austria
  - LKH Feldkirch, Interne E, Feldkirch, Vorarlberg
  - LKH Bludenz Innere Medizin, Bludenz
  - LKH Bregenz, Bregenz
  - KH Dornbirn, Innere Medizin, Dornbirn
  - Universitätsklinikum Graz, Graz
  - LKH Hohenems, Interne Intensivmedizin, Hohenems
  - Krankenhaus d. Barmherzigen Schwestern Linz, Linz
  - Universitätsklinik für Innere Medizin III mit Hämatologie, internistischer Onkologie, Infektologie, Rheumatologie und Onkologisches Zentrum, Salzburg
  - Medizinische Universität Wien, Univ.Klinik für Innere Medizin I, Abteilung für Onkologie, Vienna